CLINICAL TRIAL: NCT04540185
Title: A Phase 3, Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Polio Vaccine and NA-831 for Prophylaxis and Treatment of Early Onset of Covid-19
Brief Title: A Phase 3 Randomized Double Blind Efficacy and Safety Study of Oral Polio Vaccine and NA-831 for Covid-19
Acronym: OPV-NA831
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Biomed Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OPV-NA831
Record Dates: First submitted 2020-09-04; First posted 2020-09-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome); SARS-CoV Infection; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Poliovirus Vaccine, Oral; Drug Combinations

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Standard dose bivalent oral polio vaccine (Experimental): Biological: oral polio vaccine Bivalent OPV (GSK), 0.1 ml administered orally on a sugar lump
  Interventions: Biological: Biological: oral polio vaccine
- Comparable Placebo- 0.10 mg/kg (Placebo Comparator): Saline administered orally on a sugar lump
  Interventions: Biological: Comparable Placebo
- Standard dose of NA-831 (Experimental): Drug: neuroprotection NA-831 30 mg of NA-831in a capsule administered orally
  Interventions: Drug: NA-831
- Comparable Placebo- 30mg (Placebo Comparator): 30 mg of placebo in a capsule administered orally
  Interventions: Drug: Comparable Placebo of drug
- Standard dose of bivalent OPV and NA-831 (Experimental): Biological: oral polio vaccine Bivalent OPV (GSK), 0.1 ml administered orally on a sugar lump Plus 30 mg of neuroprotection drug NA-831 in a capsule administered orally
  Interventions: Combination Product: Combination of oral polio vaccine and NA-831
- Comparable Placebo (Placebo Comparator): Placebo of a vaccine administered orally on a sugar lump Plus 30 mg of a placebo in a capsule administered orally
  Interventions: Combination Product: Comparable Placebo of Oral Polio Vaccine and Placebo of drug

INTERVENTIONS:
Biological: Biological: oral polio vaccine — Bivalent OPV (GSK), 0.1 ml administered orally on a sugar lump
  Other Names: Oral Polio Vaccine (OPV)
  Arms: Standard dose bivalent oral polio vaccine
Biological: Comparable Placebo — Placebo of a vaccine 0.1 ml administered orally on a sugar lump
  Other Names: Placebo comparator
  Arms: Comparable Placebo- 0.10 mg/kg
Drug: NA-831 — Drug: NA-831 30 mg of NA-831 in a capsule administered orally
  Other Names: NA-81 is a neuroprotective drug
  Arms: Standard dose of NA-831
Drug: Comparable Placebo of drug — Placebo 30 mg in a capsule administered orally
  Other Names: Placebo comparator
  Arms: Comparable Placebo- 30mg
Combination Product: Combination of oral polio vaccine and NA-831 — Combination of biological: Bivalent OPV (GSK), 0.1 ml administered orally on a sugar lump and drug NA-831 30 mg in a capsule administered orally
  Other Names: OPV and Drug combination
  Arms: Standard dose of bivalent OPV and NA-831
Combination Product: Comparable Placebo of Oral Polio Vaccine and Placebo of drug — Combination of biological placebo 0.1 ml administered orally on a sugar lump and drug placebo 30 mg in a capsule administered orally
  Other Names: Placebo Comparator
  Arms: Comparable Placebo

SUMMARY:
In this randomized double blind Phase 3 clinical trial we will study the efficacy and safety of oral polio vaccine with and without NA-831 versus placebo.

DETAILED DESCRIPTION:
Early clinical studies showed that besides protecting against poliomyelitis, oral polio vaccine (OPV) reduced the number of other viruses that could be isolated from immunized children, compared with placebo recipients.

Both poliovirus and coronavirus are positive-strand RNA viruses; therefore, it is likely that they may induce and be affected by common innate immunity mechanisms. Recent reports indicate that COVID-19 may result in suppressed innate immune responses. Stimulation by live attenuated oral polio vaccines could increase resistance to infection by the causal virus, severe acute respiratory syndrome-SARS-CoV-2.

It has been discovered that SARS-CoV-2 viruses (Covid-19) can directly invade the nervous system of patients, instead of injuring the nervous system through the immune response. Increasing evidence suggests that infection with SARS-CoV-2 causes neurological deficits in a substantial proportion of affected patients. It was observed that patients surviving COVID-19 are at high risk for subsequent development of neurological disease and in particular Alzheimer's disease.

NA-831 is a new neuroprotective and neurogenesis drug that has been demonstrated its promising safety and efficacy in Phase 2A for the treatment of early onset ofAlzheimer's disease. NA-831 in oral formulation is well tolerated NA-831 with no adverse effects.

The Phase 3 clinical trial will evaluate the safety and efficacy of OPV with and without NA-831 versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are at high risk of SARS-CoV-2 infection, defined as adults whose locations or circumstances put them at appreciable risk of exposure to SARS-CoV-2 and COVID-19.
* Understands and agrees to comply with the study procedures and provides written informed consent.
* Able to comply with study procedures based on the assessment of the Investigator.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as amenorrhea for ≥12 consecutive months prior to Screening without an alternative medical cause). A follicle-stimulating hormone (FSH) level may be measured at the discretion of the Investigator to confirm postmenopausal status.
* Female participants of childbearing potential may be enrolled in the study if the participant fulfills all the following criteria:

  * Has a negative pregnancy test at Screening and on the day of the first dose (Day 1).
  * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose (Day 1).
  * Has agreed to continue adequate contraception through 3 months following the second dose on Day 29.
  * Is not currently breastfeeding.
* Male participants engaging in activity that could result in pregnancy of sexual partners must agree to practice adequate contraception and refrain from sperm donation from the time of the first dose and through 3 months after the second dose.
* Healthy adults or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.

Exclusion Criteria:

* Is acutely ill or febrile 72 hours prior to or at Screening. Fever is defined as a body temperature ≥38.0°C/100.4°F. Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled at the discretion of the Investigator.
* Is pregnant or breastfeeding.
* Known history of SARS-CoV-2 infection.
* Prior administration of an investigational coronavirus (SARS-CoV, Middle East Respiratory Syndrome [MERS]-CoV) vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19.
* Demonstrated inability to comply with the study procedures.
* An immediate family member or household member of this study's personnel.
* History of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine.
* Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
* Has received or plans to receive a vaccine within 28 days prior to the first dose (Day 1) or plans to receive a non-study vaccine within 28 days prior to or after any dose of investigational product (except for seasonal influenza vaccine).
* Has participated in an interventional clinical study within 28 days prior to the day of enrollment.
* Immunosuppressive or immunodeficient state, including human immunodeficiency virus (HIV) infection, asplenia, and recurrent severe infections.
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids ≥20 milligram (mg)/day of prednisone equivalent). Topical tacrolimus is allowed if not used within 14 days prior to Screening.
* Has received systemic immunoglobulins or blood products within 3 months prior to the day of Screening.
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a First Occurrence of COVID-19 Starting 14 Days after Second Dose of OPV with or without NA-831 | Time Frame: Day 29 (second dose) up to Day 365 (1 years after second dose)
  Number of participants infected with Covid-19 after second dose
Number of Participants with Adverse Events (AEs) or Medically Attended AEs (MAAEs) Leading to Withdrawal | Time Frame: Up to Day 365 (1 years after second dose)
  Number of participants with adverse events

SECONDARY OUTCOMES:
Number of Participants with a First Occurrence of Severe COVID-19 Starting 14 Days after Second Dose of OPV with or without NA-831 | Time Frame: Day 29 (second dose) up to Day 365 (1 years after second dose)
  Clinical signs indicative of severe COVID-19 as predefined for the study.
Number of Participants with a First Occurrence of COVID-19 Starting 14 days after Second Dose of OPV with or without NA-831 or Placebo regardless of evidence of prior SARS-CoV-2 Infection | Time Frame: Day 29 (second dose) up to Day 759 (2 years after second dose)
  Clinical signs indicative of COVID-19 and SARS-CoV-2 infection as predefined for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Tran, PhD, Study Director — Coronavirus Research Institute
Locations (10):
- United States (8):
  - Coronavirus Research Institute- Testing Site, Los Angeles, California
  - Coronavirus Research Institute, Orange, California
  - Coronavirus Research Institute-Testing Site, Palo Alto, California
  - Coronavirus Research Testing Site, San Francisco, California
  - Coronavirus Research Institute-Testing Site, Sunnyvale, California
  - Coronavirus Research Institute, Sunnyvale, California
  - Coronavirus Research Institute-Testing Site, Naperville, Illinois
  - Coronavirus Research Institute-Testing Site-, The Bronx, New York
- New Zealand (2):
  - NeuroActiva-Clinical Research Unit, Auckland
  - NeuroActiva Testing Facility of NeuroActiva (New Zealand) Ltd, Auckland

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the Study Protocol and other information if needed
Supporting Information: Study Protocol
Time Frame: 90 days after completion of the study
Access Criteria: To be verified and determined at a later date